CLINICAL TRIAL: NCT03639025
Title: The Organ Care System (OCS™) Lung Thoracic Organ Perfusion (TOP) Registry for Donor Lungs for Transplantation
Brief Title: OCS™ Lung TOP Registry For Donor Lungs for Transplantation
Acronym: TOP
Status: Active, not recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-LUN-PAS01
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Lung Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Standard Donor Lungs Primary Analysis Population: Recipients transplanted with primary analysis population eligible donor lungs preserved on the OCS™ Lung System.
  Interventions: Device: OCS Lung System
- Donor Lungs Initially Unacceptable Primary Analysis Pop.: Recipients transplanted with primary analysis population eligible donor lungs preserved on the OCS™ Lung System.
  Interventions: Device: OCS Lung System
- All Other Enrolled Patients: All OCS Lung transplanted patients that do not meet any of the above analysis populations.
  Interventions: Device: OCS Lung System

INTERVENTIONS:
Device: OCS Lung System — The OCS™ Lung System is a portable organ perfusion, ventilation, and monitoring medical device intended to preserve donor lungs in a near physiologic, ventilated, and perfused state prior to transplantation. This technology was designed to overcome the limitation of cold storage and has the potential to expand the utilization of donor lungs. The OCS™ Lung System accomplishes this by performing 3 key functions:
  * Reducing ischemic injury through the use of warm, oxygenated blood based perfusion.
  * Optimizing the lung condition by ventilatory recruitment maneuvers and high-oncotic perfusion solution supplemented with hormones and nutrients.
  * Allowing for ex-vivo functional assessment of the donor lung during preservation and prior to transplant.

SUMMARY:
Single-arm, prospective, multi-center, post-approval U.S. registry

DETAILED DESCRIPTION:
This is an all-comers registry that will enroll:

1. Patients who receive OCS™ preserved double lung transplants from either standard criteria donors or donors initially deemed unacceptable; and
2. Patients who receive a single lung transplant from OCS™ preserved lung pairs from either standard criteria donors or donors initially deemed unacceptable; and
3. All donor lungs that were perfused on OCS Lung System.

Enrolled patients will fall into one of the following three possible analysis categories:

1. TOP SCDL PAS Primary Analysis Population: will be comprised of recipients transplanted with SCDL primary analysis population eligible donor lungs preserved on the OCS™ Lung System.
2. TOP DLIDU Primary Analysis Population: Will be comprised of recipients transplanted with DLIDU primary analysis population eligible donor lungs preserved on the OCS™ Lung System.
3. All Other Enrolled Patients: will be comprised of all OCS Lung transplanted patients in the TOP Registry that do not meet any of the above analysis populations.

Patient enrollment in the TOP Registry will continue until 266 eligible DLIDU Primary Analysis Population recipients have been enrolled.

ELIGIBILITY:
This is an all-comers registry that will enroll all:

* Patients who receive OCS™ preserved double lung transplants from either standard criteria donors or donors initially deemed unacceptable; and
* Patients who receive a single lung transplant from OCS™ preserved lung pairs from either standard criteria donors or donors initially deemed unacceptable; and
* All donor lungs that were perfused on OCS Lung System.

Enrolled patients will fall into one of the following three possible analysis categories:

* TOP SCDL PAS Primary Analysis Population: will be comprised of recipients transplanted with SCDL primary analysis population eligible donor lungs preserved on the OCS™ Lung System.
* TOP DLIDU Primary Analysis Population: Will be comprised of recipients transplanted with DLIDU primary analysis population eligible donor lungs preserved on the OCS™ Lung System.
* All Other Enrolled Patients: will be comprised of all OCS Lung transplanted patients in the TOP Registry that do not meet any of the above analysis populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All lung transplant recipients whose donor lungs were preserved on the OCS™ Lung System
Sampling Method: Probability Sample
Enrollment: 458 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
12-month patient and graft survival post double-lung transplant | 12 months
  Primary Effectiveness Endpoint

SECONDARY OUTCOMES:
Standard Criteria Donor Lungs - Total ischemic time for OCS™-preserved lungs | 2 hours
  Lung ischemic time
Standard Criteria Lungs - Incidence of Primary Graft Dysfunction (PGD) grade 3 within the initial 72 hours post-transplantation (T0, T24, T48, and T72 hours) | 0, 24, 48 and 72 hours
  Primary Graft Dysfunction
Donor Lungs Initially Deemed Unacceptable - Incidence of PGD3 at 72 hours post-transplantation | 72 hours
  Primary Graft Dysfunction
Donor Lungs Initially Deemed Unacceptable - Donor Lung Utilization Rate | 1 hour
  Utilization Rate
Donor Lungs Initially Deemed Unacceptable - Incidence of PGD3 within the initial 72 hours post-transplantation | Within 72 hours post-transplantation
  Primary Graft Dysfunction

OTHER OUTCOMES:
Standard Criteria Lungs - Incidence of PGD3 at T72 hours | 72 hours
  Primary Graft Dysfunction
Total ischemia and cross-clamp times for 1st and 2nd transplanted lungs | 2 hours
  Ischemic and cross-clamp times
Kaplan-Meier patient survival estimated at Month 1, 6, 12, 24, 36, 48 and 60 | 1,6,12,24,36,48,60 months
  Survival evaluation (K-M)
Kaplan-Meier BOS-free survival estimated at Month 12, 24, 36, 48 and 60 | 12,24,36,48,60 months
  BOS free survival (K-M)
Kaplan-Meier Freedom from BOS estimated at Month 12, 24, 36, 48 and 60 | 12,24,36,48,60 months
  Freedom from BOS (K-M)
Kaplan-Meier graft survival (freedom from re-transplant/graft failure) at Month 12, 24, 36, 48 and 60 | 12,24,36,48,60 months
  Graft failure
Lung graft-related SAEs through 30 days post-transplant or discharge - Bronchial anastomotic complications; Major pulmonary-related infection | 30 days or hospital discharge (whichever is longer)
  Safety Endpoint
Survival incidence at 30 days | 30 days
  Safety Endpoint
Survival incidence at initial transplant surgery hospital discharge, if longer than 30 days. | 30 days or hospital discharge (whichever is longer)
  Safety Endpoint

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - UCSF, San Francisco, California
  - Tampa General Hospital, Tampa, Florida
  - Emory, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Nebraska Medical Center, Omaha, Nebraska
  - Duke University, Durham, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided